CLINICAL TRIAL: NCT02692235
Title: Carnitine Supplementation and Skeletal Muscle Function in Aging
Brief Title: Carnitine Supplementation and Skeletal Muscle Function
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gdansk University of Physical Education and Sport (Other)
Collaborators: National Science Centre, Poland (Other Government)
Responsible Party: Principal Investigator, Robert Olek, PhD, Gdansk University of Physical Education and Sport
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2014/15/B/NZ7/00893
Record Dates: First submitted 2016-02-13; First posted 2016-02-26 (Estimated); Results first posted 2019-05-09 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Sarcopenia
Keywords: carnitine
MeSH Terms: conditions — Sarcopenia | interventions — Carnitine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- carnitine (Experimental): 24 weeks l-carnitine-l-tartrate supplementation
  Interventions: Dietary Supplement: carnitine
- placebo (Placebo Comparator): 24 weeks isonitrogenous supplementation
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: carnitine — 1500 mg/d l-carnitine-l-tartrate
  Arms: carnitine
Dietary Supplement: placebo — isonitrogenous
  Arms: placebo

SUMMARY:
Research project objectives The primary aim of the current research project is to use carnitine supplementation as the anti-inflammatory intervention for exploring the relationship between inflammation and associated with aging reduction of skeletal muscle mass.

Hypothesis The carnitine supplementation modulates the blood cytokines concentration. Anti-inflammatory intervention delay the reduction of skeletal muscle mass associated with aging

DETAILED DESCRIPTION:
Volunteers over 65 years old (n=40) are supplemented either with carnitine or placebo for 24 weeks. Before the start, in the mid-point, and after finishing the supplementation the following primary outputs variables are performed: body composition analysis (InBody720), maximal isokinetic knee extensor peak torque (Biodex System 4 Pro), blood cytokines and carnitine concentration, blood lipid profile.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with no history of gastrointestinal disorders, cardiovascular disease or hypertension.

Exclusion Criteria:

* Subjects having any illnesses and a history of gastrointestinal disorder, cardiovascular disease, hypertension, liver and renal disease, diabetes, cancer, alcoholism or other metabolic diseases.

Ages: 65 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-02; Primary Completion 2017-03 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Olek, PhD, Principal Investigator — Gdansk University of Physical Education and Sport
Locations (1):
- University of Physical Education and Sport, Gdansk, Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 42 subjects volunteered to participate in the study. After the initial screening, 28 were included in the study (14 subject not meeting inclusion criteria) and were randomly assigned to either an L-carnitine (n=14) or a placebo supplementation group (n=14).
Period: Overall Study
Arm/Group | Carnitine | Placebo
Started | 14 | 14
Completed | 11 | 11
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Adverse Event | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carnitine | Placebo | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 14 | 14 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 14 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 28.2 (4.5) | 28.0 (5.9) | 28.1 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Blood Inflammatory Marker
Description: Serum C-reactive protein concentration determined by the enzyme immunoassay method using commercially available kit (Cloud-Clone Corp., Houston, USA)
Time Frame: baseline and after 24 weeks of supplementation period
Population: 1 male and 1 smoking female subjects excluded from the *Placebo* statistical analyses for group homogeneity
Measure: Mean (Standard Deviation); unit: mg·L^-1
Arm/Group | Carnitine | Placebo
Number analyzed (Participants) | 11 | 9
mg·L^-1
  baseline | 2.6 (0.3) | 1.8 (0.3)
  after 24 weeks | 2.9 (0.4) | 1.7 (0.3)

2. Secondary Outcome: Lipid Metabolites
Description: Change in serum lipid metabolites: total cholesterol (TCh), HDL-cholesterol (HDL), LDL-cholesterol (LDL), triglycerides (TG) determined by standard automatic analyzer Cobas 6000 (Roche Diagnostics, Mannheim, Germany)
Time Frame: baseline and after 24 weeks of supplementation period
Population: 1 male and 1 smoking female subjects excluded from the *Placebo* statistical analyses for group homogeneity
Measure: Mean (Standard Deviation); unit: mg·dL^-1
Arm/Group | Carnitine | Placebo
Number analyzed (Participants) | 11 | 9
mg·dL^-1
  TCh baseline | 233 (13) | 221 (13)
  TCh after 24 weeks | 221 (14) | 196 (14)
  HDL baseline | 69 (5) | 68 (6)
  HDL after 24 weeks | 69 (5) | 61 (3)
  LDL baseline | 140 (11) | 130 (11)
  LDL after 24 weeks | 131 (11) | 115 (13)
  TG baseline | 116 (10) | 117 (22)
  TG after 24 weeks | 105 (16) | 98 (16)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Carnitine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 1/14 | 2/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carnitine (N=14) | Placebo (N=14)
acid reflux (Gastrointestinal disorders) | 1 (1) | 1 (1)
headache and dizziness (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-02-28): https://cdn.clinicaltrials.gov/large-docs/35/NCT02692235/SAP_000.pdf
  • Study Protocol and Informed Consent Form (2015-06-22): https://cdn.clinicaltrials.gov/large-docs/35/NCT02692235/Prot_ICF_001.pdf